CLINICAL TRIAL: NCT04619069
Title: Intermittent Androgen Deprivation Therapy With or Without Stereotactic Body Radiotherapy for Molecularly Identified Hormone Sensitive Oligometastatic Prostate Cancer: A Randomized Feasibility Study
Brief Title: Intermittent Androgen Deprivation Therapy With or Without Stereotactic Body Radiotherapy for Molecularly Identified Hormone Sensitive Oligometastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iSTOP
Record Dates: First submitted 2020-10-29; First posted 2020-11-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Standard of Care (Active Comparator): Intermittent Hormone treatment (minimum of 8 months)
  Interventions: Drug: Hormone therapy
- Arm 2: SBRT to mets (Experimental): Intermittent Hormone treatment (minimum of 8 months)
  + SBRT to all sites of metastatic disease
  Interventions: Radiation: SBRT; Drug: Hormone therapy

INTERVENTIONS:
Radiation: SBRT — SBRT to all sites of metastatic disease as seen on PSMA PET scan
  Arms: Arm 2: SBRT to mets
Drug: Hormone therapy — Intermittent Hormone Therapy per physician discretion (Min. 8 months)

SUMMARY:
This study is evaluating whether adding stereotactic radiotherapy (a new, more focused type of radiotherapy) to treat all the tumours that are present will improve outcomes or not compared to drugs alone for patients who are negative on conventional imaging and positive on PSMA PET scan

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Able to provide informed consent.
3. Histologic diagnosis of prostate adenocarcinoma.
4. ECOG performance status 0-1.
5. Stage IV hormone sensitive, synchronous or metachronous oligometastatic prostate cancer as detected by PSMA PET-CT scan with no metastases visible on conventional imaging (CT chest/abdomen/pelvis and bone scan +/- MRI) performed within 3 months of starting ADT.
6. Up to a maximum of 3 PSMA avid areas of metastatic disease.
7. For patients with metachronous disease, there must be a documented PSA rise. For those who had previous prostatectomy, PSA must be > 0.2 ng/mL. For those who had previous radical radiotherapy, PSA must have risen to at least 2 ng/mL above the nadir (Phoenix definition). The primary tumor must be controlled, with no PSMA avid progression within the primary prostate.
8. All sites of disease are amenable to and can be safely treated with SBRT.

Exclusion Criteria:

1. Significant comorbidities rendering patient not suitable for ADT and/or SBRT.
2. History of malignancy within the past 5 years, excluding non-melanoma skin cancer and in-situ cancer.
3. Prior use of salvage or palliative intent ADT. Prior ADT use allowed only if it was delivered neoadjuvantly, concurrently, or adjuvantly with curative-intent treatment to the prostate or prostate bed (for patients with metachronous presentations), and at least 12 months have elapsed.
4. Castrate resistant prostate cancer.
5. Evidence of spinal cord compression.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer Patients only. Males only.
Enrollment: 60 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible patients who enroll onto the study | Through accrual completion, approx 2 years
  The primary purpose of this feasibility study is to measure the proportion of patients who are willing to enter this randomized trial

SECONDARY OUTCOMES:
Side Effects and Effectiveness | Through study completion, approx 5 years
  An important secondary purpose is to measure the side effects and effectiveness of adding stereotactic radiotherapy to all sites of disease to intermittent hormone therapy compared to intermittent hormone therapy alone, using CTCAE v.5

CONTACTS AND LOCATIONS:
Locations (1):
- Odette Cancer Centre, Toronto, Ontario, Canada